CLINICAL TRIAL: NCT04101318
Title: Investigation of a New Stoma Product for People With a Stoma
Acronym: CP288
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP288
Record Dates: First submitted 2019-09-06; First posted 2019-09-24 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-11

CONDITIONS: Peristomal Skin Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The non-Conformité Européene marked product, a Conformité Européene marked product (Experimental): Participants first received the non-Conformité Européene marked investigational product for 42±3 days. Then there was a cross-over and the participants received one of the five Conformité Européene marked comparators products, which they used the following 42±3 days.
  Interventions: Device: Non-Conformité Européene marked product; Device: Conformité Européene marked competitor products
- A Conformité Européene marked product, then the non-Conformité Européene marked product (Experimental): Participants first received one of the five Conformité Européene marked comparators products for 42±3 days. Then there was a cross-over and the participants received the non-Conformité Européene marked investigational products, which they used the following 42±3 days.
  Interventions: Device: Non-Conformité Européene marked product; Device: Conformité Européene marked competitor products

INTERVENTIONS:
Device: Non-Conformité Européene marked product — New Baseplate is not named at this point
Device: Conformité Européene marked competitor products — The Conformité Européene marked competitor products are considered Standard of Care or products considered to be part of Standard of Care in coming years.

SUMMARY:
The CP288 study is an investigation of a non-Conformité Européene marked stoma product which will be conducted in the UK, Italy, Netherlands, Germany, and Norway. The study will enroll up to 100 subjects. The study is a randomized, open-label, comparative study.

DETAILED DESCRIPTION:
Enrolled participant with an ileostomy or colostomy with liquid output were randomized to test either the non-Conformité Européene marked investigational product or one of the five comparators Conformité Européene marked products first and then will be crossed over to receive the opposite intervention.

The participant will first be included in an information and inclusion visit (V0) and after signing all consent forms will complete three test visits (V1, V2, and V3). Each participant will be enrolled for 2 × 42±3 days in total for the entire investigation, thus for a maximum of 90 days.

The study is a randomised, controlled, open-label, comparative, cross-over, multicentre investigation with two test periods. The study was conducted in four different countries (UK, Germany, Italy, and Norway) with a total of six sites participating.

The study is now complete.

ELIGIBILITY:
Inclusion Criteria:

1. Has given informed consent to participate by signing the informed consent signature form.
2. Has an ileostomy or colostomy with liquid output (defined by a 6-7 on the Bristol Scale)
3. Currently using a flat product
4. Be at least 18 years of age and have full legal capacity
5. Have had their stoma for at least three months (90 days)
6. Can use a product with a max cut size of 40 mm
7. Has experienced leakage* under the baseplate at least three times within the last 14 days. *leakage defined as output seeping under the baseplate (Appendix 6 - Classification of leakage)
8. Has symptoms of peristomal skin complications or has peristomal skin complications defined by at least one of the below

   1. Has experienced symptoms of skin complications (itching, burning, pain) within the last fourteen days
   2. Has experienced red skin in the inner circle (within three cm from stoma edge) within the last fourteen days
   3. Has skin complication (assessed by Principal Investigator, or delegate) in the inner circle (within three cm from stoma edge) of the peristomal area
9. Is able to handle the electronic diary (questionnaire/ photo) themselves.
10. Is able to handle (apply, remove, cut etc.) the product themselves
11. Is willing to not use barrier film or barrier cream during the investigation
12. Is willing and suitable (determined by Principal Investigator, or delegate) to use a flat custom cut one-piece open or a two-piece open product during the investigation.
13. Is willing to change the product (1pc) or baseplate (2pc) at least every fourth days.

Exclusion Criteria:

1. Is currently receiving or have within the past 60 days received radio-and/or chemotherapy

   - low doses chemotherapy (assessed by Principal Investigator) is allowed for indications other than cancer.
2. Is currently receiving or have within the past month received topical steroid treatment in the peristomal skin area, e.g. lotion or spray.

   * Low dose systemic steroid treatment (e.g. inhalation) assessed by the Principal Investigator are allowed.
   * Other systemic steroid treatment (e.g. injection, or tablet) are not allowed.
3. Is breastfeeding
4. Is pregnant (based on pregnancy test -urine)
5. Has known hypersensitivity towards any of the products used in the investigation

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazarena Mazzarro, MD, Study Director — Coloplast A/S
Locations (1):
- Ragene Saetre, Larvik, Norway

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 79 participants were recruited from six sites across four countries (UK, Germany, Italy, and Norway) and encompassed the safety population.
Pre-assignment Details: 79 recruited participants were randomized. Of those 7 participants were excluded as two participants wanted to be discontinued, one participant had device deficiency leading to an Adverse event, two participants had device deficiency not leading to an Adverse event, one participant had an adverse event, and one participant was discontinued due to other reasons.
  So 72 participants constituted the intention to treat (ITT) population.
Groups:
- The Non-Conformité Européene Marked Product, Then a Conformité Européene Marked Product: Participants first received the non-Conformité Européene marked investigational product for 42±3 days. Then there was a cross-over and the participants received one of the five Conformité Européene marked comparators products, which they used the following 42±3 days.
Period: First Intervention (42 +/- 3 Days)
Arm/Group | The Non-Conformité Européene Marked Product, Then a Conformité Européene Marked Product | A Conformité Européene Marked Product, Then the Non-Conformité Européene Marked Product
Started | 34 | 38
Received Allocated Intervention | 34 | 36
Completed | 34 | 36
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention (42 +/- 3 Days)
Arm/Group | The Non-Conformité Européene Marked Product, Then a Conformité Européene Marked Product | A Conformité Européene Marked Product, Then the Non-Conformité Européene Marked Product
Started | 34 | 36
Received Allocated Intervention | 33 | 35
Completed | 33 | 35
Not Completed | 1 | 1
Not completed — Device deficiency not leading to an adverse event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population Baseline Measures: Arm 1: Participants first received the non-Conformité Européene marked investigational product for 42±3 days. Then there was a cross-over and the participants received one of the five Conformité Européene marked comparators products, which they used the following 42±3 days.
  Arm 2: Participants first received one of the five Conformité Européene marked comparators products for 42±3 days. Then there was a cross-over and the participants received the non-Conformité Européene marked investigational products, which they used the following 42±3 days.
Arm/Group | Total ITT Population Baseline Measures
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 13
  Germany | 35
  Italy | 2
  United Kingdom | 22
Weight (kg) [Mean (Standard Deviation); unit: kg] | 80.5 (21.0)
Height (cm) [Mean (Standard Deviation); unit: cm] | 170.4 (11.3)
BMI (kg/cm^2) [Mean (Standard Deviation); unit: kg/cm^2] | 27.6 (6.3)
Stoma age [Mean (Standard Deviation); unit: years] | 11.2 (10.9)
Type of stoma [Count of Participants; unit: Participants]
  Colostomy | 15
  Ileostomy | 57

OUTCOME MEASURES:

1. Primary Outcome: Max Itching Within a Week at Steady State
Description: Participant were asked to rate their itching around the ostomy on a scale of 0-10 with 0= no itch ad 10= worst possible peristomal skin itch. The primary outcome measure was done on the Intended to Treat population. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within a week at steady state
Population: The intention to treat population (full analysis set) was constituted by all randomized subjects with a valid informed consent who have been exposed to at least one product, and with valid information on at least one product with respect to the endpoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Non-Conformité Européene Marked Investigational Baseplate Change: The assessment was done after a baseplate change with the non-Conformité Européene marked investigational product
- Conformité Européene Marked Comparator Baseplate Change: The assessment was done after a baseplate change with one of the five Conformité Européene marked comparator products
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
score on a scale | 2.5 [2.0 to 3.0] | 2.4 [1.9 to 2.9]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.625, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Model was with the following fixed effects: product and period. Subject and the interaction between product and subject were random effects; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.38 to 0.62] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

2. Secondary Outcome: Percentage of Participants With Varying Frequency of Itching Skin in the Past 14 Days by End of Treatment
Description: Participants were asked how often they had experienced itchy skin around their ostomy in the past 14 days by the end of treatment. The data was distributed into five categories: "None of the time", "A little of the time", Some of the time", A lot of the time", and "All of the time". The results are shown as the percentages of answers for that category out of a total of a 100% (comprising the total of all answers from all the categories). When adding the number for each of the five categories it sums up to 100. So the results are shown as "how many percentages are the answers from one category out of a total of 100% (all the answers)?".
Time Frame: past 14 days by end of treatment
Population: The intention to treat population (full analysis set) was constituted by all randomized subjects with a valid informed consent who have been exposed to at least one product, and with valid information on at least one product with respect to the endpoints. The Outcome Measure Data Table depict (seen below) the percentages of total from the statistical data model analyzing 67 participants with measurements in at least one of the arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 58 | 60
percentage of participants
  None of the time | 22 | 22
  A little of the time | 37 | 22
  Some of the time | 25 | 29
  A lot of the time | 16 | 24
  All of the time | 0 | 3
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.036, Proportional odds ratio model — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Ordinal regression model for itching evaluated on a 5 point scale. Product and period are fixed effects and subject is a random effect; Odds Ratio (OR) = 1.737, 95% CI 2-sided [1.038 to 2.908] — Odds ratio, marginal= Arm1/Arm2

3. Secondary Outcome: Max Pain Within a Week at Steady State
Description: Participant were asked to rate their pain around the ostomy on a scale of 0-10 with 0= no pain ad 10= worst possible pain. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
score on a scale | 1.4 [0.9 to 1.9] | 1.7 [1.3 to 2.2]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.202, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; The mode had following fixed effects: product and period. Subject and the interaction between product and subject were random effects; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.90 to 0.20] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

4. Secondary Outcome: Percentage of Participants With Varying Frequency of Pain in the Past 14 Days by End of Treatment
Description: Participants were asked how often they had experienced pain around their ostomy in the past 14 days by the end of treatment. The data was distributed into five categories: "None of the time", "A little of the time", Some of the time", A lot of the time", and "All of the time". The results are shown as the percentages of answers for that category out of a total of a 100% (comprising the total of all answers from all the categories). When adding the number for each of the five categories it sums up to 100. So the results are shown as "how many percentages are the answers from one category out of a total of 100% (all the answers)?".
Time Frame: past 14 days by end of treatment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 58 | 60
percentage of participants
  None of the time | 45 | 43
  A little of the time | 39 | 33
  Some of the time | 10 | 20
  A lot of the time | 6 | 4
  All of the time | 0 | 0
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.267, Proportional odds ratio model — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Ordinal regression model for pain evaluated on a 5 point scale. Product and period are fixed effects and subject is a random effect; Odds Ratio (OR) = 1.369, 95% CI 2-sided [0.781 to 2.401] — Odds ratio, marginal= Arm1/Arm2

5. Secondary Outcome: Max Burning Within a Week at Steady State
Description: Participant were asked to rate burning around the ostomy on a scale of 0-10 with 0= no itch ad 10= worst possible burning sensation. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
score on a scale | 1.8 [1.3 to 2.3] | 2.0 [1.5 to 2.5]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.545, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.57 to 0.30] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

6. Secondary Outcome: Percentage of Participants With Varying Frequency of Burning in the Past 14 Days by End of Treatment
Description: Participants were asked how often they had experienced a burning sensation around their ostomy in the past 14 days by the end of treatment. The data was distributed into five categories: "None of the time", "A little of the time", Some of the time", A lot of the time", and "All of the time". The results are shown as the percentages of answers for that category out of a total of a 100% (comprising the total of all answers from all the categories). When adding the number for each of the five categories it sums up to 100. So the results are shown as "how many percentages are the answers from one category out of a total of 100% (all the answers)?".
Time Frame: past 14 days by end of treatment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 58 | 60
percentage of participants
  None of the time | 37 | 39
  A little of the time | 39 | 27
  Some of the time | 16 | 22
  A lot of the time | 8 | 10
  All of the time | 0 | 2
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.293, Proportional odds ratio model — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Ordinal regression model for burning evaluated on a 5 point scale. Product and period are fixed effects and subject is a random effect; Odds Ratio (OR) = 1.316, 95% CI 2-sided [0.783 to 2.211] — Odds ratio, marginal= Arm1/Arm2

7. Secondary Outcome: Bleeding Around the Ostomy at Each Baseplate Change at Steady State
Description: Participant were asked if they had experienced bleeding around the ostomy within 1 week. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Mean odds, marginal
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
Mean odds, marginal | 0.38 [0.27 to 0.52] | 0.46 [0.34 to 0.62]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; There is no difference between the two arms; Test type: Superiority; p = 0.375, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; generalized linear mixed repeated model with fixed effects; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.53 to 1.27] — Odds ratio, marginal= Arm1/Arm2

8. Secondary Outcome: Weeping Around the Ostomy at Each Baseplate Change at Steady State
Description: Participant were asked if they had experienced weeping around the ostomy within 1 week. Steady state period of the treatment period begins after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Mean odds, marginal
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
Mean odds, marginal | 0.38 [0.26 to 0.56] | 0.46 [0.32 to 0.65]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.482, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; generalized linear mixed repeated model with fixed effects; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.49 to 1.40] — Odds ratio, marginal= Arm1/Arm2

9. Secondary Outcome: Ulcers Around the Ostomy at Each Baseplate Change at Steady State
Description: Participant were asked if they had experienced ulcers around the ostomy within 1 week. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Mean odds, marginal
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
Mean odds, marginal | 0.40 [0.27 to 0.58] | 0.57 [0.41 to 0.80]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.151, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; generalized linear mixed repeated model with fixed effects; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.43 to 1.14]; Odds ratio, marginal= Arm1/Arm2

10. Secondary Outcome: Max Overall Physical Discomfort Within a Week Per Baseplate Change at Steady State
Description: Participant were asked to rate their overall physical discomfort around the ostomy on a scale of 0-10 with 0= no discomfort/difficulty and 10= a lot of discomfort/difficulty. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- CE Marked Comparator Baseplate Change: The assessment was done after a baseplate change with one of the five CE marked comparator products
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | CE Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
score on a scale | 1.9 [1.4 to 2.4] | 1.8 [1.3 to 2.3]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs CE Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.725, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.39 to 0.56] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

11. Secondary Outcome: Max Overall Ability to Move Around Within a Week Per Baseplate Change at Steady State
Description: Participant were asked to rate their overall ability to move around on a scale of 0-10 with 0= no discomfort/difficulty and 10= a lot of discomfort/difficulty. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
score on a scale | 1.3 [0.9 to 1.8] | 1.3 [0.8 to 1.7]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.721, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.39 to 0.56] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

12. Secondary Outcome: Max Overall Ability to Stick the Stoma Bag Adhesive to the Skin Within a Week Per Baseplate Change at Steady State
Description: Participant were asked to rate the overall ability to stick the stoma bag adhesive to their skin since last change of product on a scale of 0-10 with 0= no discomfort/difficulty and 10= a lot of discomfort/difficulty. Steady state period of the treatment period began after three weeks of product use.
Time Frame: Within one week at steady state
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
score on a scale | 0.8 [0.4 to 1.2] | 0.9 [0.5 to 1.3]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.753, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.38 to 0.28] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

13. Secondary Outcome: Discoloration Area (cm^2) Per Baseplate Change at Steady State
Description: Participant were asked to take photos of their peristomal skin at each baseplate change. The discoloration area of the peristomal skin was determined using an algorithm. The algorithm estimated the area of the discolored skin (divided into three different zones). Steady state period of the treatment period began after three weeks of product use.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
cm^2 | 18.5 [15.4 to 21.7] | 17.2 [14.1 to 20.3]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.331, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.37, 95% CI 2-sided [-1.43 to 4.18] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

14. Secondary Outcome: Intensity of Discolorated Area Scored Per Baseplate Change at Steady State After Three Weeks of Product Use
Description: Photos of the peristomal skin was taken at each baseplate change. The intensity was determined with an overlay to the artificial intelligence algorithm. The overlay divided the area into ten different intensity intervals: "Intensity interval 1"=0-10 …., "Intensity interval 10"=91-100% redness. The score was then calculated as follows: 1*(Interval 1 measurement)..+ 10*(Interval 10 measurement). Thus, if the area was within the first interval (0-10% redness) it was multiplied with 1 or within Interval 10 it was multiplied with 10, resulting in a intensity score for the total area. If there is no discoloration the score is 0, and there is no theoretical maximum. A large score equals a high intensity on the skin. In the description of the endpoint (appendix. 1 in CIP), it was to be determined in the inner and outer zone per baseplate change at steady state. However, the algorithm only estimated a total intensity score; thus, the intensity will not be reported per inner and outer zone.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Total intensity area score (cm^2)
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 59 | 65
Total intensity area score (cm^2) | 107.1 [84.6 to 129.5] | 95.4 [73.4 to 117.3]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.239, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.68, 95% CI 2-sided [-7.98 to 31.34] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

15. Secondary Outcome: Total Discoloration, Erosion, and Tissue Overgrowth (DET) Score by End of Treatment at Steady State
Description: Participant were asked to take photos close to the stoma, which was then assessed by a sponsor or health care professionals. They determined the discoloration, erosion, and tissue overgrowth domain by scoring the area (0-3, with 3 being a large area affected), and severity (1-2, with 2 being the highest severity) affected by each domain. Each three domains contributes to the calculation of the total Discoloration, Erosion and Tissue overgrowth score (DET) going from a scale of 0 to 15 ("Normal skin" (DET=0), "Mild" (DET=2- 3), "Moderate" (DET=4- 6), and "Severe" (7-15)).
  Steady state period of the treatment period began after three weeks of product use.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 69 | 70
score on a scale | 3.5 [2.9 to 4.2] | 3.8 [3.2 to 4.5]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.322, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Model was with the following fixed effects: product and period. Subject was a random effect; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.91 to 0.31] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

16. Secondary Outcome: Discoloration Item Score by End of Treatment at Steady State
Description: Participant were asked to take photos close to the stoma, which was then assessed by a sponsor or health care professionals. Discoloration is a part of the discoloration, erosion, and tissue overgrowth (DET) score where all domains are assess to give a total DET score, with a min of 0 and max of 15. The discoloration domain was scored by area (0-3, with 3 being a large area affected), and severity (1-2, with 2 being the highest severity) affected and the scores were added together for a total discoloration score (with the max total score being 5). The area is assessed first and if this is 0 then the score for discoloration is 0, meaning the severity is not assessed. This means that the maximum score possible is 5 and the lowest score possible is 0 and the higher the score the more discolored skin.
  Steady state period of the treatment period began after three weeks of product use
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 69 | 70
score on a scale | 2.4 [2.1 to 2.8] | 2.6 [2.3 to 2.9]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.343, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Model was with the following fixed effects: product and period. Subject was a random effect; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.44 to 0.15] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

17. Secondary Outcome: Erosion Item Score by End of Treatment at Steady State
Description: Participant were asked to take photos close to the stoma, which was then assessed by a sponsor or health care professionals. Erosion is a part of the discoloration, erosion, and tissue overgrowth (DET) score where all domains are assess to give a total DET score, with a min of 0 and max of 15.The erosion domain was determined by scoring the area (0-3, with 3 being a large area affected), and severity (1-2, with 2 being the highest severity) affected and then adding the scores together for a total score (with the max total score being 5). The area is assessed first and if this is 0 then the score for erosion is 0, meaning the severity is not assessed. This means that the maximum score possible is 5 and the lowest score possible is 0 and the higher the score the more eroded skin.
  Steady state period of the treatment period began after three weeks of product use.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 69 | 70
score on a scale | 0.7 [0.4 to 1.0] | 0.9 [0.6 to 1.2]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.387, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Model was with the following fixed effects: product and period. Subject was a random effect; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.53 to 0.21] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

18. Secondary Outcome: Tissue Overgrowth Item Score by End of Treatment at Steady State
Description: Participant were asked to take photos close to the stoma, which was then assessed by a sponsor or health care professionals. Tissue overgrowth is a part of the discoloration, erosion, and tissue overgrowth (DET) score where all domains are assess to give a total DET score, with a min of 0 and max of 15. The Tissue Overgrowth domain was assessed by scoring the area (0-3, with 3 being a large area affected), and severity (1-2, with 2 being the highest severity) affected and then adding the scores together for a total score (with the max total score being 5). The area is assessed first and if this is 0 then the score for tissue overgrowth is 0, meaning the severity is not assessed. This means that the maximum score possible is 5 and the lowest score possible is 0 and the higher the score the more tissue overgrowth.
  Steady state period of the treatment period began after three weeks of product use.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Non-Conformité Européene Marked Investigational Baseplate Change | Conformité Européene Marked Comparator Baseplate Change
Number analyzed (Participants) | 69 | 70
score on a scale | 0.3 [0.1 to 0.6] | 0.3 [0.1 to 0.6]
Statistical Analysis 1: Comparison: Non-Conformité Européene Marked Investigational Baseplate Change vs Conformité Européene Marked Comparator Baseplate Change; Null hypothesis: There is no difference between the two arms; Test type: Superiority; p = 0.899, Mixed Models Analysis — The threshold for statistical significance was p=0.05. Furthermore, p-value was not adjusted for multiple comparisons; Model was with the following fixed effects: product and period. Subject was a random effect; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.18 to 0.16] — Difference between Arm 1 and Arm 2= Mean (Arm 1) - Mean (Arm 2)

ADVERSE EVENTS:
Time Frame: Each subject was enrolled for 2 x 42±3 days in total for the entire investigation, thus for a maximum of 90 days.
Description: The relationship to the investigational or comparator product were collected. The Safety population constituted the subjects who have given informed consent and were 79 participants.
  The participants in each arm represent an adverse event reported that was either: "Not related", "Unlikely related", "Possibly related", "Probably related", or "Definitely related", to the Non-Conformité Européene Marked Product or the Conformité Européene Marked product.
Groups:
- Non-Conformité Européene Marked Product: Product is not named at this point
- Conformité Européene Marked Products: 1-piece and 2-piece stoma devices already on the market.
- Total Safety Population: This arm/group constitutes the safety population
Arm/Group | Non-Conformité Européene Marked Product | Conformité Européene Marked Products | Total Safety Population
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/73 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/73 | 5/79
Other Adverse Events (participants affected / at risk) | 27/74 | 28/73 | 43/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Conformité Européene Marked Product (N=74) | Conformité Européene Marked Products (N=73) | Total Safety Population (N=79)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Ileus: patient experienced severe pan in the stomach.
Exacerbated cystic fibrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Heart attack (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Guillain-barre syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Feeding line infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Conformité Européene Marked Product (N=74) | Conformité Européene Marked Products (N=73) | Total Safety Population (N=79)
Dental abscess (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hay fever (General disorders) | 0 (0) | 0 (0) | 2 (2)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tiredness (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2)
Diarrohea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Leakage and bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Bleeding from stoma (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Frequent watery stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Output more liquid than normal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
One bladder at stoma (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Swollen stoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Painful/Sore Throat (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Excessive sweating (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — EXCESSIVE SWEATING (REPORTED FEELING HOT - TEMPERATURE 37.4 DEGREES CELSIUS)
Prexia (38.1 DEGREES C) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 4 (6)
Muscle cramps in legs (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bleeding skin (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (7) | 6 (10)
Blotchy skin around stoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Broken skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Burning around stoma (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (3)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Allergic contact dermatitis
Cuts under stoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dark patches of skin around stoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dry/flaky skin around stoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erosions/Ulcers (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Pain (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (10) | 11 (17)
Itching skin (Skin and subcutaneous tissue disorders) | 12 (13) | 8 (12) | 19 (25)
Redness (Skin and subcutaneous tissue disorders) | 9 (11) | 9 (14) | 12 (22)
Stinging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (4) | 7 (8) | 9 (12)
Skin complication (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (3)
Leakage and skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Oozing skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT04101318/Prot_SAP_000.pdf